CLINICAL TRIAL: NCT04461886
Title: A Long-term Study of NPC-12G Gel in Neurofibromatosis Type I
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-12G-5
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Neurofibromatosis
MeSH Terms: conditions — Neurofibromatoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NPC-12G gel (Experimental): NPC-12G gel is containing 0.2% Sirolimus
  Interventions: Drug: NPC-12G gel

INTERVENTIONS:
Drug: NPC-12G gel — NPC-12G gel is containing 0.2% Sirolimus

SUMMARY:
The purpose of this tria is to evaluate the safety and efficacy of long-term treatment with NPC-12G gel to patients with neurofibromatosis type I.

DETAILED DESCRIPTION:
A Phase 3, open-label, uncontrolled, multicenter study to evaluate the safety and efficacy of long-term treatment with NPC-12G gel for patients with neurofibromatosis type I. Patients who meet all entry criteria for this trial apply NPC-12G gel twice a day for 52 weeks or more. Approximately 100 eligible patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as neurofibromatosis type 1 based on the clinical diagnostic criteria in guideline of Japanese Dermatological Association
2. Patients participated in a Phase II/III investigator-initiated clinical trial for neurofibromatosis type I (OSD-001-004) who wish to continue treatment of the investigational drug
3. At the time of enrollment, patients who are able to choose ten evaluable target lesions for efficacy (at least 5)..
4. Patients who have evaluable skin neurofibromas at baseline.
5. Males and females who are 3 years old or elder at the time of informed consent.
6. Patients who (or whose guardian) give a written informed consent in understanding and willingness after having received enough explanation regarding the study participation.
7. Patients whose use or continued use of the investigational drug is judged to be reasonable by the principal investigator or sub-investigator.

Exclusion Criteria:

1. Patients who occurred serious adverse effects, who discontinued the sudy due to adverse effects, or who discontinued the trial due to withdrew of their consent in the Phase II/III investigator-initiated study of neurofibromatosis type I (OSD-001-004)
2. Patients with abnormal findings (e.g., pneumonia) in the results of chest x-ray at the time of screening
3. Patients with creatinine clearance of less than 50 mL/min
4. Patients with poorly controlled dyslipidemia (serum triglycerides >500 mg/dL or LDL cholesterol >190 mg/dL even with treatment)
5. Patients who have complications such as infection, cardiac, hepatic, pulmonary, renal, or hematological diseases and malignant tumors that are considered unsuitable for participation in this trial.
6. Patients with alcohol sensitivity or allergy to an ingredient of the study drug (Sirolimus)
7. Female patients who are pregnant, may be pregnant, or are lactating
8. Patients (including male patients with a fertile partner) who cannot consent to use adequate contraception from the date of consent to 12 weeks after the end of treatment
9. Patients who participated in any other clinical trial or clinical study, other than the OSD-001-004 study, and have taken an investigational or investigational drug within 6 months prior to the date of the consent
10. Patients who are participating in an observational study during this trial
11. Patients who are considered by the investigator as unsuitable for participation in this trial

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Discontinuation rate associated with adverse events (Kaplan-Meier method) | 52 weeks
  Number of Adverse events leading to discontinuation

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Osaka University Hospital, Suita-shi, Osaka
  - Jikei University Hospital, Minato-ku, Tokyo
  - Fukuoka University Hospital, Fukuoka
  - Tottori University Hospital, Tottori

IPD SHARING:
Plan to Share IPD: Undecided